CLINICAL TRIAL: NCT04683146
Title: Effectiveness of Pre-surgical Hand Washing in Reducing Bacterial Load, Using an Alcoholic Solution of Chlorhexidine Digluconate and Potassium Sorbate
Brief Title: Pre-surgical Antisepsis Using an Alcoholic Solution of Chlorhexidine Digluconate and Potassium Sorbate ( Sorbectol )
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centro Ortopedico y Quirurgico del Pie (Other)
Responsible Party: Principal Investigator, Ricardo Becerro de Bengoa Vallejo, Principal investigator, Centro Ortopedico y Quirurgico del Pie
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RICBEC2
Record Dates: First submitted 2020-12-20; First posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Antisepsis
MeSH Terms: interventions — Ethanol; chlorhexidine gluconate; Sorbic Acid

STUDY DESIGN:
Intervention Model Description: Crossover Assignment Crossover design is used
Who Masked: Outcomes Assessor
Masking Description: The samples will be sent to the laboratory with numbers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hand antisepsis with propanolol-1 60% (Active Comparator): Effectiveness of pre-surgical hand washing in reducing bacterial load using propranolol- 1 60% as control.
  Interventions: Drug: Hand antisepsis with Propanolol- 1 60%.; Drug: Hand antisepsis with a solution of alcohol, chlorhexidine digluconate and potassium sorbate.
- Hand antisepsis with solution of alcohol, chlorhexidine digluconate and potassium sorbate (Active Comparator): Effectiveness of pre-surgical hand washing in reducing bacterial load using a solution of alcohol, chlorhexidine digluconate and potassium sorbate
  Interventions: Drug: Hand antisepsis with Propanolol- 1 60%.; Drug: Hand antisepsis with a solution of alcohol, chlorhexidine digluconate and potassium sorbate.

INTERVENTIONS:
Drug: Hand antisepsis with Propanolol- 1 60%. — * Pre-washing for one minute with neutral soap to remove the transient flora.
  * Hand antisepsis using Propanolol-1 60% in both hands.
  * Bacterial sample collection from right hand.
  * Sterile surgical glove in both hands.
  * Bacterial sample collection from left hand three hours later
Drug: Hand antisepsis with a solution of alcohol, chlorhexidine digluconate and potassium sorbate. — * Pre-washing for one minute with neutral soap to remove the transient flora.
  * Hand antisepsis using a solution of alcohol, chlorhexidine digluconate and potassium sorbate.
  * Bacterial sample collection from right hand.
  * Sterile surgical glove in both hands.
  * Bacterial sample collection from left hand three hours later.

SUMMARY:
The present study evaluates the effects of bactericidal load reduction after surgical hand antisepsis using the reference antiseptic product propanol- 1 60% as control versus a surgical hand antisepsis with addition of a solution of alcohol, chlorhexidine digluconate and potassium sorbate in order to test if pass the standard european norm 12791.

DETAILED DESCRIPTION:
The investigators conducted a crossover clinical trial to evaluate the antiseptic effectiveness of surgical hand antisepsis using propan-ol-1 60% by using the reference antiseptic product propan-ol-1 60% as control versus a surgical hand antisepsis with addition of a solution of alcohol, chlorhexidine digluconate and potassium sorbate in order to test if pass the standard european norm 12791. Samples will be taken from the hands of each volunteer after a surgical hands antiseptic.

ELIGIBILITY:
Inclusion Criteria:

* Participants with healthy skin in both hands and short fingernails.
* No use of antibacterial agents for at least three days before the intervention.
* Not received antibiotic treatment for at least ten days before the intervention.

Exclusion Criteria:

* Known systemic pathologies
* Wearing hand jewelry on the hands
* Allergy to any ingredient of which the solutions used in the clinical trial are composed
* Cognitive and / or motor limitation that makes it impossible to carry out instructions for hand washing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-03-10 (Estimated); Primary Completion 2021-03-24 (Estimated); Study Completion 2021-06-05 (Estimated)

PRIMARY OUTCOMES:
Reduction of bacterial load immediately after hand scrub | Change from bacterial load at 5 minutes]
  Participants will scrub the antiseptic solution vigorously from hand to the wrists according with the standard handrub procedure

SECONDARY OUTCOMES:
Reduction of bacterial load after 3 hours of hand scrub | Change from bacterial load at 3 hours
  Participants will scrub the antiseptic solution vigorously from hand to the wrists according with the standard handrub procedure after 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Becerro de Bengoa Vallejo, Principal Investigator — Universidad Complutense de Madrid

IPD SHARING:
Plan to Share IPD: No
A number will be assigned to each participant